CLINICAL TRIAL: NCT01839097
Title: Phase 1 Dose Finding Study of Belinostat Plus Cyclophosphamide/Vincristine/Doxorubicin/Prednisone (CHOP) Regimen (BelCHOP) for Treatment of Patients With Peripheral T-cell Lymphoma(PTCL)
Brief Title: Phase 1 Dose Finding Study of Belinostat for Treatment of Patients With Peripheral T-cell Lymphoma (PTCL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acrotech Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPI-BEL-12-104
Record Dates: First submitted 2013-04-09; First posted 2013-04-24 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Peripheral T-cell Lymphoma
Keywords: PTCL; Maximum Tolerated Dose; Belinostat
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — belinostat; Cyclophosphamide; Vincristine; Doxorubicin; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dose Finding Phase (Experimental): This is a Phase 1 dose finding study using the traditional escalation rule of 3+3 design to evaluate the Maximum Tolerated Dose of Belinostat when administered in combination with CHOP. In Part A of the study, up to three sequential dose cohorts will enroll a maximum of 6 patients each.
  Enrollment will begin with the enrollment of patients into Cohort 3.
  On Day 1 of each 21-day treatment cycle, the study treatment will start with belinostat followed by CHOP regimen.
  Interventions: Drug: Belinostat; Drug: CHOP

INTERVENTIONS:
Drug: Belinostat — Belinostat will be administered by intravenous infusion once daily for up to 5 days depending on the dose cohort as follows:
  * Cohort 1: belinostat 1000 mg/m2 IV on Day 1
  * Cohort 2: belinostat 1000 mg/m2 IV on Day 1-2
  * Cohort 3: belinostat 1000 mg/m2 IV on Day 1-3
  * Cohort 4: belinostat 1000 mg/m2 IV on Day 1-4
  * Cohort 5: belinostat 1000 mg/m2 IV on Day 1-5
  Other Names: PXD101
Drug: CHOP — Cyclophosphamide - 750 mg/m2 - IV - Day 1
  Vincristine - 1.4 mg/m2 - IV - Day 1
  Doxorubicin - 50mg/m2 - IV - Day 1
  Prednisone 100mg PO - On Day 1 Prednisone will be administered after chemotherapy part of CHOP, and on Day 2-5 after belinostat.
  Other Names: Cyclophosphamide; Vincristine; Doxorubicin; Prednisone

SUMMARY:
The primary objective of this study is to determine the Maximum Tolerated Dose (MTD) for belinostat when combined with CHOP regimen and establish the recommended belinostat dose for the Phase 3 study.

DETAILED DESCRIPTION:
This is a Phase 1 dose finding study using the traditional escalation rule of 3+3 design to evaluate the Maximum Tolerated Dose (MTD) of belinostat when administered in combination with CHOP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Life Expectancy > 3 months
* Histologically confirmed diagnosis of PTCL
* Patients with transformed CTCL eligible for CHOP regimen
* Measurable disease based on Cheson 2007 criteria
* Eastern Cooperative Oncology Group (ECOG) performance status < 2

Exclusion Criteria:

* Known active Hepatitis B/ Hepatitis C/ HIV infection
* Known, uncontrolled CNS metastases or primary CNS lymphoma
* Deep vein thrombosis diagnosed within 3 months
* Ongoing treatment for pre-existing cardiovascular disease
* Neuropathy Grade 3 or more
* Previous extensive radiotherapy except limited field RT for locally advanced nasal NK PTCL or for pain palliation
* Prior therapy with severely myelotoxic regimens, including autologous and allogenic stem cell transplantation
* Prior therapy with HDAC inhibitors (except for CTCL)
* Inadequate hematological, hepatic, or renal function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | up to 5 days
  To determine the MTD for belinostat when combined with CHOP regimen and establish the Phase 3 recommended belinostat dose.

SECONDARY OUTCOMES:
Safety and tolerance | up to 5 days
  To assess safety and tolerance of belinostat when given in combination with CHOP regimen. Safety and tolerance will be mainly characterized by the number and severity of treatment emergent adverse events, and treatment related AEs that occur or worsen after the first dose of study treatment.
Overall Response Rate | 126 days
  Overall response rate (ORR) after 6 cycles of BelCHOP regimen
Effectiveness of study drug | 126 days
  Pharmacokinetics of belinostat when co-administered with CHOP regimen. The concentration of Belinostat to assess the effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Mi Rim Choi, MD, Study Director — Spectrum Pharmaceuticals, Inc
Locations (8):
- United States (8):
  - Yale University, New Haven, Connecticut
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Hematology - Oncology Associates of Northern NJ P.A, Morristown, New Jersey
  - Columbia University Medical Center/Center for Lymphiod Malignancies, New York, New York
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Derived] Johnston PB, Cashen AF, Nikolinakos PG, Beaven AW, Barta SK, Bhat G, Hasal SJ, De Vos S, Oki Y, Deng C, Foss FM. Belinostat in combination with standard cyclophosphamide, doxorubicin, vincristine and prednisone as first-line treatment for patients with newly diagnosed peripheral T-cell lymphoma. Exp Hematol Oncol. 2021 Feb 18;10(1):15. doi: 10.1186/s40164-021-00203-8. PMID 33602316